## STUDY PROTOCOL

Prospective Monitoring of Non-Vitamin K Oral Anticoagulants in Older Adults with Atrial Fibrillation and Frailty

**Preparation or Update Date:** 

04/05/2021

# **Protocol Revision Summary**

Date

# **Summary of Changes**

04/05/2021

Protocol preparation for study registration

#### **BACKGROUND**

- 1. Non-vitamin K antagonist oral anticoagulants (NOACs) dabigatran, rivaroxaban, apixaban, and edoxaban for treatment of atrial fibrillation (AF)
  - a. Dabigatran Approved October 19, 2010 (1)

RE-LY Trial (Dabigatran vs Warfarin)

- i. N=18,113, follow-up: 2.0y
- ii. Composite event of stroke/non-CNS systemic embolism: 1.5%/y vs 1.7%/y (HR: 0.66; 95% CI: 0.53-0.82)
- iii. Safety endpoints: Major bleeding: 2.7%/y vs 3.4%/y (HR: 0.93; 95% CI: 0.81-1.07)
- b. Rivaroxaban Approved July 1, 2011(2)

ROCKET-AF Trial (Rivaroxaban vs Warfarin) (3)

- i. N=14,264, Follow-up: 1.9y
- ii. Composite event of stroke/non-CNS systemic embolism: 1.7%/y vs 2.2%/y (HR: 0.79; 95% CI: 0.66-0.96)
- iii. Safety endpoints: Major bleeding: 3.6%/y vs 3.4%/y (HR: 1.04; 95% CI: 0.90-1.20)
- c. Apixaban Approved December 28, 2012 (4)

ARISTOTLE (Apixaban vs Warfarin) (5)

- i. N=18,201, Follow-up: 1.8y
- ii. Composite event of stroke/non-CNS systemic embolism: 1.3%/y vs 1.6%/y (HR: 0.79; 95% CI: 0.66-0.95)
- iii. Safety endpoints: Major bleeding: 2.1%/y vs 3.1%/y (HR: 0.69; 95% CI: 0.60-0.80)
- d. Edoxaban Approved January 18, 2015 (6)

ENGAGE AF-TIMI (Edoxaban vs Warfarin) (7)

- i. N=21,105, Follow-up: 2.8y
- ii. Composite event of stroke/non-CNS systemic embolism: 1.2%/y vs 1.5%/y (HR: 0.79; 95% CI: 0.63-0.99)
- iii. Safety endpoints: Major bleeding: 2.8%/y vs 3.4%/y (HR: 0.80; 95% CI: 0.71-0.91)
- 2. Summary of 2019 ACC/AHA/ESC Guidelines for management of atrial fibrillation (8)
  - a. For patients with AF and an elevated CHA2DS2-VASc score of 2 or greater in men or 3 or greater in women, oral anticoagulants are recommended (Level of Evidence: A to B-R).

- b. NOACs (dabigatran, rivaroxaban, apixaban, and edoxaban) are recommended over warfarin in NOAC-eligible patients with AF (except with moderate-to-severe mitral stenosis or a mechanical heart valve) (Level of Evidence: A).
- c. In patients with AF (except with moderate-to-severe mitral stenosis or a mechanical heart valve), the CHA2DS2-VASc score is recommended for assessment of stroke risk (Level of Evidence: B).
- d. In patients with AF, anticoagulant therapy should be individualized on the basis of shared decision-making after discussion of the absolute risks and relative risks of stroke and bleeding, as well as the patient's values and preferences (Level of Evidence: C).
- e. For patients with AF (except with moderate- to-severe mitral stenosis or a mechanical heart valve) and a CHA2DS2-VASc score of 0 in men or 1 in women, it is reasonable to omit anticoagulant therapy (Level of Evidence: B).
- f. For patients with AF who have a CHA2DS2-VASc score of 2 or greater in men or 3 or greater in women and who have end-stage chronic kidney disease (CKD; creatinine clearance [CrCl] <15 mL/min) or are on dialysis, it might be reasonable to prescribe warfarin (INR 2.0 to 3.0) or apixaban for oral anticoagulation (Level of Evidence: B-NR).
- g. For patients with AF (except with moderate- to-severe mitral stenosis or a mechanical heart valve) and moderate-to-severe CKD (serum creatinine ≥1.5 mg/dL [apixaban], CrCl 15 to 30 mL/min [dabigatran], CrCl ≤50 mL/min [rivaroxaban], or CrCl 15 to 50 mL/ min [edoxaban]) with an elevated CHA2DS2- VASc score, treatment with reduced doses of direct thrombin or factor Xa inhibitors may be considered (eg, dabigatran, rivaroxaban, apixaban, or edoxaban) (Level of Evidence: B-R).
- h. For patients with AF (except with moderate- to-severe mitral stenosis or a mechanical heart valve) and a CHA2DS2-VASc score of 1 in men and 2 in women, prescribing an oral anticoagulant to reduce thromboembolic stroke risk may be considered (Level of evidence: C-LD).

#### STUDY OVERVIEW AND DESIGN

- 1. Study aims: To emulate a prospective surveillance of the effectiveness and safety of NOACs vs a comparator (warfarin) in older adults with Atrial Fibrillation and different frailty status.
- 2. Data source(s):
  - a. Commercial data Optum and MarketScan (2010-latest data available)

- b. Medicare data (2013-latest data available)
- 3. Study design (see Figure 1): The monitoring analysis will include 1) retrospective analysis of available data (2013-2018) at the time of first analysis (March 2021) and 2) prospective analysis of new data (2019-2020) as they become available to the researchers. Within each database and by frailty status (frail vs non-frail), we will emulate annual updating of data by creating a propensity score (PS)-matched cohort of new users every 1-year interval. Each sequential cohort will be followed for development of the outcomes of interest. At the end of each interval, time-to-event data from all sequential cohorts will be pooled for outcome analysis. The surveillance will be performed by frailty status (frail vs non-frail) at the time of drug initiation.

Figure 1. Schematic of sequential monitoring design



### STUDY POPULATION

- 1. Study population (see Figure 2) is created <u>for each calendar interval and by frailty status for each NOAC</u> vs warfarin comparison.
- 2. Initiation of NOAC or comparator (warfarin)
  - a. NOAC: any of dabigatran, rivaroxaban, apixaban, edoxaban
  - b. Index date (day 0): prescription fill from July 1, 2013
- 3. Assessment of eligibility (eligibility assessment window: [-183, 0] days) See Appendix for list of codes. If a patient meets the eligibility criteria more than once, only the first record will be included.

- a. Continuous enrollment in medical and drug insurance (up to 30-day gap allowed; no HMO in Medicare data)
- b. Diagnosis of AF (CCW definition; outpatient diagnosis x2 or inpatient x1)
- c. CHA2DS2-VASc score ≥2 (moderate or high risk for stroke)
- d. No prior use of NOAC or warfarin (exposure wash-out window: [-183, -1] days)
- e. No recent hospitalization for stroke or major bleeding (outcome wash-out window: [-60, 0] days)
- f. No recent nursing facility stay: [-60, 0] days
  - i. Place of service: 31 (skilled nursing facility), 32 (nursing facility), 33 (custodial care facility)
  - CPT codes: 99301, 99302, 99303, 99311, 99312, 99313, 99315, 99316, 99379,
     99380, G0066
- g. Excluded if age <65 years or exposure to both drugs on day 0
- h. Contraindication to either drug (exclusion assessment window: [-183, 0] days)
  - i. Valvular heart disease or mechanical heart valve
  - ii. Intracranial or retroperitoneal hemorrhage
  - iii. Chronic kidney disease stage V, end-stage renal disease, or dialysis
  - iv. Other indications for anticoagulation therapy (venous thromboembolism or joint replacement)

Figure 2. Study design outline for comparative effectiveness and safety analysis



#### **MEASUREMENTS**

- 1. Exposure to NOAC or comparator (each NOAC analyzed separately)
  - a. NOAC: dabigatran, rivaroxaban, apixaban, or edoxaban
  - b. Warfarin (comparator)
  - c. Exposure risk window and gap between treatments allowed: 3 days (primary analysis) or 5 days (sensitivity analysis)

#### 2. Outcomes

- a. Effectiveness endpoints:
  - i. a composite of stroke or systemic embolism (primary)
- b. Safety endpoints:
  - i. Major bleeding (primary)
  - ii. All-cause mortality

### 3. Covariates

- a. Sociodemographic information: age, sex, race, dual eligibility (for Medicare data)
- b. Diseases: Chronic Conditions Data Warehouse (CCW) chronic conditions (see Table 2), provided in the Medicare Beneficiary Summary File (first date of satisfying the claims-based algorithm for individual conditions is available; considered present if this date is earlier than the index date)
- c. Fall history: any fall diagnosis codes
- d. Prescription drugs: selected ATC3 classes (chosen based on prevalence in a representative Medicare population)
- e. CHA2DS2-VASc score
- f. HAS-BLED score (9)
- g. Gagne combined comorbidity score (10)
- h. Claims-based frailty index (11): Frailty status will be defined as non-frail if <0.20 or frail if ≥0.20
- i. Health care utilization: number of hospitalization days calculated from inpatient dataset; number of skilled nursing facility days calculated from skilled nursing facility dataset

## **Table 2. CCW Chronic Conditions (12)**

| Acquired Hypothyroidism | Chronic Kidney Disease |
|---|---|
| Acute Myocardial Infarction | Chronic Obstructive Pulmonary Disease |
| Alzheimer's Disease, Related Disorders, or Senile<br>Dementia | Depression |
| Anemia | Diabetes |
| Asthma | Glaucoma |
| Heart failure | Hip / Pelvic Fracture |
| Benign Prostatic Hyperplasia | Hyperlipidemia |
| | Hypertension |
| Cancer (any of the following): Cancer, Colorectal | Ischemic Heart Disease |
| Cancer, Endometrial Cancer, Breast | Osteoporosis |
| Cancer, Lung Cancer, Prostate | Rheumatoid Arthritis / Osteoarthritis |
| Cancer, 1 rostate | Stroke / Transient Ischemic Attack |
| Cataract | |

## STATISTICAL ANALYSIS

### Estimation of treatment effectiveness and safety within each database

- 1. Monitoring framework: Monitoring framework: We will emulate annual updating of data by dividing each database for each NOAC-warfarin comparison into consecutive 1-year intervals. The monitoring begins on July 1, 2013-December 31, 2014, and 1-year intervals afterwards. Within each interval, we will fit a propensity score (PS) model and find PS-matched pairs. As new data become available every year, we will identify additional PS-matched pairs. Each sequential cohort will be followed for development of the outcomes of interest. At the end of each interval, time-to-event data from all sequential cohorts will be analyzed. The surveillance will be performed by frailty status at the time of drug initiation. The signal for effectiveness and safety will be determined using the maximized sequential probability ratio test. (13)
- 2. PS analysis: PS model will be estimated by frailty status (frail vs non-frail) within each cohort. We will use logistic regression that estimates the probability of receiving the drug of interest as a function

of sociodemographic characteristics, diseases, prescription drugs, comorbidity index, frailty index, CHA2DS2-VASc score, HAS-BLED score, and indicators for each 1-year interval. We will perform a 1:1 ratio nearest-neighbor PS matching, with a caliper of 0.2 of the standard deviation of the logit PS (Austin et al. Pharm Stat. 2011;10:150-61). We will evaluate balance in covariates using standard mean difference (<0.1 is considered adequate balance) within each surveillance cohort.

- 3. Primary analysis for effectiveness and safety: We will estimate the rate difference and 95% confidence interval (CI) of the effectiveness and safety endpoints by frailty status (frail vs non-frail). We will also use Cox proportional hazards regression to estimate the hazard ratios (HR) and 95% CI by frailty status (frail vs non-frail). The follow-up will begin on day 1 and end on the day of development of the effectiveness or safety endpoints or the earliest of the following censoring events: switching or discontinuation of the study drug, death not due to the outcome of interest, disenrollment, and end of data period (see Figure 1). Proportional hazards assumptions will be checked using Schoenfeld residuals.
- 4. Subgroup analyses for primary endpoints:
  - a. Age (65-74 years vs  $\geq$ 75 years)
  - b. Sex
  - c. Race (Black vs non-Black)
  - d. Major multimorbidity burden/pattern (informed by latent class analysis)
  - e. Dementia (CCW definition)
  - f. Fall history
  - g. CHA2DS2-VASc (≥4 vs 2-3)
  - h. HAS-BLED ( $\geq 2$  or  $\leq 2$ )
- 5. Sensitivity analysis for primary effectiveness and safety endpoints:
  - a. "intention-to-treat" analysis with a maximum follow-up time of 1 year from the index date
  - b. Exposure risk window or grace period of 5 days

## Estimation of the pooled treatment effectiveness and safety

The treatment effect estimates from 3 databases will be combined using meta-analysis techniques.
 We will examine the heterogeneity of treatment effect using Cochrane Q statistics and I-square statistics. If there is no statistically significant evidence of treatment effect heterogeneity, we will use

inverse probability fixed-effects model to pool the database-specific estimates. If there is significant treatment effect heterogeneity, we will use random-effects model.

2. Reporting of prospective monitoring results: When a statistically significant signal is detected from the pooled analysis for the primary endpoints of effectiveness or safety from pre-specified interim analysis or at the end of the data period (12/31/2020), the findings will be reported.

#### REFERENCES

- Boehringer Ingelheim Pharmaceuticals, Inc. PRADAXA (dabigatran etexilate mesylat) [package insert]. U.S. Food and Drug Administration website.
   https://www.accessdata.fda.gov/drugsatfda\_docs/label/2010/022512s000lbl.pdf. Revised October 2010. Accessed Feb 22, 2021.
- Janssen Pharmaceuticals, Inc. XARELTO (rivaroxaban) [package insert]. U.S. Food and Drug Administration website.
   <a href="https://www.accessdata.fda.gov/drugsatfda\_docs/label/2011/022406s000lbl.pdf">https://www.accessdata.fda.gov/drugsatfda\_docs/label/2011/022406s000lbl.pdf</a>. Revised July 2011. Accessed Feb 22, 2021.
- 3. Patel MR, Mahaffey KW, Garg J, Pan G, Singer DE, Hacke W, et al. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. N Engl J Med. 2011;365(10):883-91.
- 4. Bristol-Myers Squibb Co. ELIQUIS (apixaban) [package insert]. U.S. Food and Drug Administration website. <a href="https://www.accessdata.fda.gov/drugsatfda\_docs/label/2012/202155s000lbl.pdf">https://www.accessdata.fda.gov/drugsatfda\_docs/label/2012/202155s000lbl.pdf</a>. Revised December 2012. Accessed Feb 22, 2021.
- 5. Granger CB, Alexander JH, McMurray JJ, Lopes RD, Hylek EM, Hanna M, et al. Apixaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2011;365(11):981-92.
- 6. Daiichi Sankyo, Inc. SAVAYSA (edoxaban) [package insert]. U.S. Food and Drug Administration website.<a href="https://www.accessdata.fda.gov/drugsatfda\_docs/label/2015/206316lbl.pdf">https://www.accessdata.fda.gov/drugsatfda\_docs/label/2015/206316lbl.pdf</a>. Revised January 2015. Accessed May 20, 2019.
- 7. Giugliano RP, Ruff CT, Braunwald E, Murphy SA, Wiviott SD, Halperin JL, et al. Edoxaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2013;369(22):2093-104.
- 8. January CT, Wann LS, Calkins H, Chen LY, Cigarroa JE, Cleveland JC, Jr., et al. 2019 AHA/ACC/HRS Focused Update of the 2014 AHA/ACC/HRS Guideline for the Management of Patients With Atrial Fibrillation: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society in Collaboration With the Society of Thoracic Surgeons. Circulation. 2019;140(2):e125-e51.
- 9. Pisters R, Lane DA, Nieuwlaat R, de Vos CB, Crijns HJ, Lip GY. A novel user-friendly score (HAS-BLED) to assess 1-year risk of major bleeding in patients with atrial fibrillation: the Euro Heart Survey. Chest. 2010;138(5):1093-100.
- 10. Combined Comorbidity Score for Claims Data [Internet]. Available from: <a href="https://www.drugepi.org/dope/software">https://www.drugepi.org/dope/software</a>.
- 11. Claims-Based Frailty Index [Internet]. 2020 [cited December 1, 2020]. Available from: <a href="https://dataverse.harvard.edu/dataverse/cfi/">https://dataverse.harvard.edu/dataverse/cfi/</a>.

- 12. Chronic Conditions Data Warehouse [Internet]. 2020. Available from: <a href="https://www2.ccwdata.org/web/guest/condition-categories/">https://www2.ccwdata.org/web/guest/condition-categories/</a>.
- 13. Brown JS, Kulldorff M, Chan KA, Davis RL, Graham D, Pettus PT, et al. Early detection of adverse drug events within population-based health networks: application of sequential testing methods. Pharmacoepidemiol Drug Saf. 2007;16(12):1275-84.

### **APPENDIX**

# **ATC Drug Class**

A02B DRUGS FOR PEPTIC ULCER AND GASTRO-OESOPHAGEAL REFLUX DISEASE (GORD)

A06A DRUGS FOR CONSTIPATION

A10A INSULINS AND ANALOGUES

A10B BLOOD GLUCOSE LOWERING DRUGS, EXCL. INSULINS

A11 VITAMINS

A12B POTASSIUM SUPPLEMENTS

**B01A ANTITHROMBOTIC AGENTS** 

**B02A ANTIFIBRINOLYTICS** 

**B02B VITAMIN K AND OTHER HEMOSTATICS** 

**B03A IRON ANTIANEMIC PREPARATIONS** 

B03B VITAMIN B12 AND FOLIC ACID

B03X OTHER ANTIANEMIC PREPARATIONS in ATC

**B05A BLOOD AND RELATED PRODUCTS** 

B05B IV solutions used in parenteral administration of fluids, electrolytes and nutrients

C01A CARDIAC GLYCOSIDES

C01B ANTIARRHYTHMICS, CLASS I AND III

C01C CARDIAC STIMULANTS EXCL. CARDIAC GLYCOSIDES

C01D VASODILATORS USED IN CARDIAC DISEASES

C02D ARTERIOLAR SMOOTH MUSCLE, AGENTS ACTING ON

C03A LOW-CEILING DIURETICS, THIAZIDES

C03C HIGH-CEILING DIURETICS

C03D POTASSIUM-SPARING DIURETICS

C07 beta-Adrenergic Blocking Agents

C08C SELECTIVE CALCIUM CHANNEL BLOCKERS WITH MAINLY VASCULAR EFFECTS

C08D SELECTIVE CALCIUM CHANNEL BLOCKERS WITH DIRECT CARDIAC EFFECTS

C09A ACE INHIBITORS, PLAIN

C09B ACE INHIBITORS, COMBINATIONS

C09C ANGIOTENSIN II RECEPTOR BLOCKERS (ARBs), PLAIN

C09D ANGIOTENSIN II RECEPTOR BLOCKERS (ARBs), COMBINATIONS

C09X OTHER AGENTS ACTING ON THE RENIN-ANGIOTENSIN SYSTEM in ATC

C10A LIPID MODIFYING AGENTS, PLAIN

D03 PREPARATIONS FOR TREATMENT OF WOUNDS AND ULCERS

**G04B UROLOGICALS** 

G04C DRUGS USED IN BENIGN PROSTATIC HYPERTROPHY

 ${\tt H02A\ CORTICOSTEROIDS\ FOR\ SYSTEMIC\ USE,\ PLAIN}$ 

H03A THYROID PREPARATIONS

J01 ANTIBACTERIALS FOR SYSTEMIC USE

J02 ANTIMYCOTICS FOR SYSTEMIC USE

J05 ANTIVIRALS FOR SYSTEMIC USE

J07 VACCINES

L01 ANTINEOPLASTIC AGENTS

L02 ENDOCRINE THERAPY ANTINEOPLASTIC AND IMMUNOMODULATING AGENTS

L03 IMMUNOSTIMULANTS

L04 IMMUNOSUPPRESSANTS

M01A ANTIINFLAMMATORY AND ANTIRHEUMATIC PRODUCTS, NON-STEROIDS

M03B MUSCLE RELAXANTS, CENTRALLY ACTING AGENTS

M04A ANTIGOUT PREPARATIONS

M05B DRUGS AFFECTING BONE STRUCTURE AND MINERALIZATION

N02A OPIOID ANALGESICS

N02B OTHER ANALGESICS AND ANTIPYRETICS in ATC

N03A ANTIEPILEPTICS

N04 ANTI-PARKINSON DRUGS

N05A ANTIPSYCHOTICS

N05B ANXIOLYTICS

N05C HYPNOTICS AND SEDATIVES

N06A ANTIDEPRESSANTS

N06B PSYCHOSTIMULANTS, AGENTS USED FOR ADHD AND NOOTROPICS

N06D ANTI-DEMENTIA DRUGS

**R03A ADRENERGICS, INHALANTS** 

R03B OTHER DRUGS FOR OBSTRUCTIVE AIRWAY DISEASES, INHALANTS in ATC

**R03C ADRENERGICS FOR SYSTEMIC USE** 

R03D OTHER SYSTEMIC DRUGS FOR OBSTRUCTIVE AIRWAY DISEASES in ATC

R06A ANTIHISTAMINES FOR SYSTEMIC USE

S01E ANTIGLAUCOMA PREPARATIONS AND MIOTICS

## **Covariate and Outcome Codes**

### Valvular Heart Disease/Mechanical Heart Valve


# CKD5, ESRD, or Dialysis


| ICD10PX | 5A1.D80Z | Performance of Urinary Filtration, 6-18 hrs/day |
|---------|----------|-------------------------------------------------|
| ICD10PX | 5A1.D90Z | Performance of Urinary Filtration, >18 hrs/day |

# Venous Thromboembolism


# Joint Replacement


| ICD10PX 0SR.9029 Replace R Hip Jt w Metal on Poly, Cement, Open | |
|---|---|
| ICD10PX 0SR.902A Replace R Hip Jt w Metal on Poly, Uncement, Open | |
| ICD10PX 0SR.902Z Replacement of R Hip Jt with Metal on Poly, Open Appro | oach |
| ICD10PX 0SR.9039 Replacement of R Hip Jt with Ceramic, Cement, Open Ap | |
| ICD10PX 0SR.903A Replace of R Hip Jt with Ceramic, Uncement, Open Appr | - |
| ICD10PX 0SR.903Z Replacement of Right Hip Joint with Ceramic, Open App | |
| ICD10PX 0SR.9049 Replace R Hip Jt w Ceramic on Poly, Cement, Open | |
| ICD10PX 0SR.904A Replace R Hip Jt w Ceramic on Poly, Uncement, Open | |
| ICD10PX 0SR.904Z Replacement of R Hip Jt with Ceramic on Poly, Open Ap | proach |
| ICD10PX 0SR.9069 Replace of R Hip Jt with Zirc on Poly, Cement, Open App | • |
| ICD10PX 0SR.906A Replace R Hip Jt w Zirc on Poly, Uncement, Open | , |
| ICD10PX 0SR.906Z Replacement of R Hip Jt with Zirc on Poly, Open Approa | ch |
| ICD10PX 0SR.907Z Replacement of Right Hip Joint with Autol Sub, Open Ap | |
| ICD10PX 0SR.90EZ Replacement of Right Hip Joint with Artc Spcr, Open Ap | - |
| ICD10PX 0SR.90J9 Replace of R Hip Jt with Synth Sub, Cement, Open Appro | - |
| ICD10PX 0SR.90JA Replace of R Hip Jt with Synth Sub, Uncement, Open Ap | |
| ICD10PX 0SR.90JZ Replacement of Right Hip Joint with Synth Sub, Open Ap | • |
| ICD10PX 0SR.90KZ Replacement of R Hip Jt with Nonaut Sub, Open Approach | _ |
| ICD10PX 0SR.A009 Replace R Hip Jt, Acetab w Polyeth, Cement, Open | |
| ICD10PX 0SR.A00A Replace R Hip Jt, Acetab w Polyeth, Uncement, Open | |
| ICD10PX 0SR.A00Z Replacement of R Hip Jt, Acetab with Polyeth, Open App | roach |
| ICD10PX 0SR.A019 Replace R Hip Jt, Acetab w Metal, Cement, Open | |
| ICD10PX 0SR.A01A Replace R Hip Jt, Acetab w Metal, Uncement, Open | |
| ICD10PX 0SR.A01Z Replacement of R Hip Jt, Acetab with Metal, Open Appro | oach |
| ICD10PX 0SR.A039 Replace R Hip Jt, Acetab w Ceramic, Cement, Open | |
| ICD10PX 0SR.A03A Replace R Hip Jt, Acetab w Ceramic, Uncement, Open | |
| ICD10PX 0SR.A03Z Replacement of R Hip Jt, Acetab with Ceramic, Open Ap | proach |
| ICD10PX 0SR.A07Z Replace of R Hip Jt, Acetab with Autol Sub, Open Appro | |
| ICD10PX 0SR.A0J9 Replace R Hip Jt, Acetab w Synth Sub, Cement, Open | |
| ICD10PX 0SR.A0JA Replace R Hip Jt, Acetab w Synth Sub, Uncement, Open | |
| ICD10PX 0SR.A0JZ Replace of R Hip Jt, Acetab with Synth Sub, Open Appro | ach |
| ICD10PX 0SR.A0KZ Replace of R Hip Jt, Acetab with Nonaut Sub, Open Appr | roach |
| ICD10PX 0SR.B019 Replacement of L Hip Jt with Metal, Cement, Open Appr | oach |
| ICD10PX 0SR.B01A Replacement of L Hip Jt with Metal, Uncement, Open Ap | proach |
| ICD10PX 0SR.B01Z Replacement of Left Hip Joint with Metal, Open Approach | h |
| ICD10PX 0SR.B029 Replace L Hip Jt w Metal on Poly, Cement, Open | |
| ICD10PX 0SR.B02A Replace L Hip Jt w Metal on Poly, Uncement, Open | |
| ICD10PX 0SR.B02Z Replacement of L Hip Jt with Metal on Poly, Open Appro | oach |
| ICD10PX 0SR.B039 Replacement of L Hip Jt with Ceramic, Cement, Open Ap | proach |
| ICD10PX 0SR.B03A Replace of L Hip Jt with Ceramic, Uncernent, Open Appr | oach |
| ICD10PX 0SR.B03Z Replacement of Left Hip Joint with Ceramic, Open Appro | oach |
| ICD10PX 0SR.B049 Replace L Hip Jt w Ceramic on Poly, Cement, Open | |
| ICD10DV OCD DOAA Doules LIE LOCK DILLIE | |
| ICD10PX 0SR.B04A Replace L Hip Jt w Ceramic on Poly, Uncement, Open | |
| ICD10PX 0SR.B04A Replace L Hip Jt w Ceramic on Poly, Uncement, Open ICD10PX 0SR.B04Z Replacement of L Hip Jt with Ceramic on Poly, Open Ap | proach |


## **Falls**


```
ICD10DX
                W05.1XXD Fall from non-moving nonmotorized scooter, subs enentr
ICD10DX
                W05.1XXS Fall from non-moving nonmotorized scooter, sequela
ICD10DX
                W05.2
                            Fall from non-moving motorized mobility scooter
ICD10DX
                W05.2XXA Fall from non-moving motorized mobility scooter, init enentr
ICD10DX
                W05.2XXD Fall from non-moving motorized mobility scooter, subs enentr
ICD10DX
                W05.2XXS Fall from non-moving motorized mobility scooter, sequela
ICD10DX
                W06
                            Fall from bed
ICD10DX
                W06.XXXA Fall from bed, initial encounter
ICD10DX
                W06.XXXD Fall from bed, subsequent encounter
ICD10DX
                W06.XXXS Fall from bed, sequela
ICD10DX
                W07
                            Fall from chair
                W07.XXXA Fall from chair, initial encounter
ICD10DX
ICD10DX
                W07.XXXD Fall from chair, subsequent encounter
ICD10DX
                W07.XXXS Fall from chair, sequela
                W08
ICD10DX
                            Fall from other furniture
ICD10DX
                W08.XXXA Fall from other furniture, initial encounter
ICD10DX
                W08.XXXD Fall from other furniture, subsequent encounter
ICD10DX
                W08.XXXS Fall from other furniture, sequela
ICD10DX
                W10
                            Fall on and from stairs and steps
ICD10DX
                W10.0
                            Fall (on)(from) escalator
ICD10DX
                W10.0XXA Fall (on)(from) escalator, initial encounter
ICD10DX
                W10.0XXD Fall (on)(from) escalator, subsequent encounter
ICD10DX
                W10.0XXS Fall (on)(from) escalator, sequela
ICD10DX
                W10.1
                            Fall (on)(from) sidewalk curb
ICD10DX
                W10.1XXA Fall (on)(from) sidewalk curb, initial encounter
ICD10DX
                W10.1XXD Fall (on)(from) sidewalk curb, subsequent encounter
ICD10DX
                W10.1XXS Fall (on)(from) sidewalk curb, sequela
                W10.2
ICD10DX
                            Fall (on)(from) incline
ICD10DX
                W10.2XXA Fall (on)(from) incline, initial encounter
ICD10DX
                W10.2XXD Fall (on)(from) incline, subsequent encounter
ICD10DX
                W10.2XXS Fall (on)(from) incline, sequela
ICD10DX
                W10.8
                            Fall (on) (from) other stairs and steps
ICD10DX
                W10.8XXA Fall (on) (from) other stairs and steps, initial encounter
ICD10DX
                W10.8XXD Fall (on) (from) other stairs and steps, subs encntr
ICD10DX
                W10.8XXS Fall (on) (from) other stairs and steps, sequela
ICD10DX
                W10.9
                            Fall (on) (from) unspecified stairs and steps
ICD10DX
                W10.9XXA Fall (on) (from) unspecified stairs and steps, init enentr
ICD10DX
                W10.9XXD Fall (on) (from) unspecified stairs and steps, subs encntr
ICD10DX
                W10.9XXS Fall (on) (from) unspecified stairs and steps, sequela
ICD10DX
                W18.1
                            Fall from or off toilet
ICD10DX
                W18.11
                            Fall from or off toilet w/o strike against object
ICD10DX
                W18.11XA Fall from or off toilet w/o strike against object, init
ICD10DX
                W18.11XD Fall from or off toilet w/o strike against object, subs
ICD10DX
                W18.11XS Fall from or off toilet w/o strike against object, sequela
                            Fall from or off toilet w subsequent striking against object
ICD10DX
                W18.12
```


# **Ischemic Stroke**


# Systemic Embolism


## **Critical Site Bleeding**


#### **Intracranial Bleeding**

SOURCE CODE DESCRIPTION


## **Retroperitoneal Bleeding**


## **Non-critical Site Bleeding**


# **GI Bleeding**


#### Transfusion

